CLINICAL TRIAL: NCT03825913
Title: Feasibility and Safety Profile of a 3-month Aerobic and Resistance Exercise Intervention for Individuals Diagnosed With Melanoma
Brief Title: 3-month Aerobic and Resistance Exercise Intervention for Individuals Diagnosed With Melanoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: two key faculty members are no longer part of the study and institution
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Eduard Tiozzo, PhD, Instructor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20180174
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Active Comparator): Subjects in the exercise group will participate in a 3-month exercise program at the University of Miami UHealth Fitness and Wellness Center. Participants will complete two exercise sessions a week, each 45-60 minutes long and on a one-on-one basis.
  In addition to two site visits, the participants will receive a tailored daily home-based walking plan. The participants will use physical activity trackers (Fitbit®), with an ultimate goal of achieving 10,000 steps by the end of the intervention.
  Participants in the exercise intervention will complete 24 sessions.
  Interventions: Behavioral: Exercise Intervention
- Wellness Intervention (Sham Comparator): For 3 months, the wellness education group will not be offered any form of supervised exercise program or receive any specific instructions on physical activity as part of the study. The participants in this group will attend educational sessions about different wellness topics, such as nutrition, sleep, weight management, mindfulness, and the overall benefits of increased physical activity. The wellness visits will be held two times per month, and similar to the exercise sessions of the intervention arm, they will be 45-60 minutes long and on a one-on-one basis. Participants in the wellness education group will complete 6 sessions.
  Interventions: Behavioral: Wellness Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Training sessions will include a split routine based on the day of the week.
  * Session 1 (e.g. Tuesday) - aerobic exercise (20-30 min) followed by resistance training (10 stacked-weight machines: leg press, leg extension, leg curl, chest press, latissimus pull, shoulder press, seated row, triceps press, biceps curl, and chest fly) for 1-2 sets of 8-12 repetitions.
  * Session 2 (e.g. Thursday) - resistance bands and body weight exercises (4-6 exercises, 2 sets of 10-20 repetitions) followed by core exercises (2-3 sets of 10-20 repetitions) and aerobic training (20-30 min) at the end.
  The starting training intensities will be at 50-55% of each individual's estimated maximum heart rate for aerobic exercise and one-repetition maximum for resistance training (assessed at baseline only for chest press and leg press). We plan a 5% monthly increase in the intensity to reach 65-70%% of one's maximum efforts by the end of the intervention.
  Arms: Exercise Intervention
Behavioral: Wellness Intervention — In our setting, ten lectures in nutrition, exercise and various complementary and integrative medicine topics (e.g. acupuncture and Chinese medicine, mindfulness, quality sleep, etc.) were implemented among non-cancer individuals and modified based on their feedback.
  Arms: Wellness Intervention

SUMMARY:
Our proposed study will focus on addressing the feasibility, safety and benefits of a 3-month exercise intervention among individuals diagnosed with melanoma.

The study will be conducted at University of Miami Miller School of Medicine. Eligible participants (n=24) will be randomized into 3 months of wellness education (n=12) or structured exercise (n=12).

DETAILED DESCRIPTION:
Our proposed study will focus on addressing the feasibility, safety and benefits of a 3-month exercise intervention among individuals diagnosed with melanoma.

The study will be conducted at University of Miami Miller School of Medicine. The eligible participants will meet the following inclusion and exclusion criteria.

Inclusion criteria: (a) men and women (≥ 18 years of age) with melanoma cancer within one year from diagnosis, (b) not meeting the guidelines for physical activity (less than 150 minutes of moderate intensity activity or 75 minutes of vigorous intensity activity a week for 6 weeks prior the enrollment) (c) a commitment to two weekly supervised exercise sessions or bi-monthly educational sessions for three months at University of Miami Miller School of Medicine and (d) able to understand, read and write English.

Exclusion criteria: (a) participants for whom physical activity is contraindicated because of comorbid conditions, (b) participants with dementia, altered mental status or psychiatric condition and (c) participants who are unwilling or unable to provide informed consent.

The participants (n=24) will be randomized into 3 months of: 1) wellness education (n=12) or 2) structured exercise (n=12). All participants will receive standard treatment as directed by their oncologists. Individuals in the wellness education group will attend bi-monthly sessions where they will receive general wellness information pertaining to physical activity, nutrition, sleep, weight management and mindfulness. Individuals in the structured exercise group will attend supervised exercise sessions twice per week and receive a tailored daily walking plan using physical activity trackers. A comprehensive assessment will be conducted at baseline and 3-months, which will include demographics, medical and treatment history, anthropometrics, quality of life, physical fitness, past and current sun exposure, fatigue, and nutritional status. We plan the following specific aims:

Aim 1: To assess feasibility, adherence, and safety of a 3-month supervised exercise program in melanoma patients.

Aim 2: To evaluate the impact of a 3-month supervised exercise program on quality of life in melanoma patients.

Aim 3: To evaluate the effect of a 3-month supervised exercise program on cardiorespiratory fitness and muscular strength in melanoma patients.

ELIGIBILITY:
Inclusion criteria: (a) men and women (≥ 18 years of age) with a diagnosis of melanoma cancer within one year from diagnosis, (b) not meeting the guidelines for physical activity (less than 150 minutes of moderate intensity activity or 75 minutes of vigorous intensity activity a week for 6 weeks prior the enrollment) (c) a commitment to two weekly supervised exercise sessions or bi-monthly educational sessions for three months at University of Miami Miller School of Medicine (d) and able to understand, read and write English.

Exclusion criteria: (a) participants for whom physical activity is contraindicated because of comorbid conditions, (b) participants with dementia, altered mental status or psychiatric condition and (c) participants who are unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Feasibility Assessment | 12 weeks
  Less than 20% attrition rate for the intervention group
Adherence Assessment | 12 weeks
  80% or higher of the exercise sessions completed

SECONDARY OUTCOMES:
FACT-M (Functional Assessment of Cancer Therapy - Melanoma) | 6 and 12 weeks
  Quality of Life
6-minute Walk Test | 12 weeks
  Cardiorespiratory Fitness
Hand Grip | 12 weeks
  Muscular Strength
30-sec Chair Stand | 12 weeks
  Functional Status
Food Frequency Questionnaire | 12 weeks
  Nutritional Intake
SEBI (Sun Exposure and Behavior Inventory) | 12 weeks
  Sun Exposure
FACIT (Functional Assessment of Chronic Illness Therapy | 6 and 12 weeks
  Fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Tiozzo, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No